CLINICAL TRIAL: NCT05005676
Title: Evaluation of the New Three-dimensional Acceleromyograph TOF 3D Compared With the Established TOF Watch SX.
Brief Title: Evaluation of the New Acceleromyograph TOF 3D
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kreiskrankenhaus Dormagen (Other)
Responsible Party: Principal Investigator, Stefan Soltesz, Prof. Dr. Stefan Soltesz, Kreiskrankenhaus Dormagen
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: TOF 3D
Record Dates: First submitted 2021-08-02; First posted 2021-08-13 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Assessment of a New Acceleromyograph; Neuromuscular Block

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- adductor pollicis AP (Experimental): Measurement site: M.adductor pollicis of both arms.
  Interventions: Diagnostic Test: acceleromyography
- Corrugator supercilii CS (Experimental): Measurement site: M. corrugator supercilii at both sides
  Interventions: Diagnostic Test: acceleromyography

INTERVENTIONS:
Diagnostic Test: acceleromyography — Simultaneous measurement of the time course of a neuromuscular block with 2 acceleromyographs

SUMMARY:
The TOF 3D is a new acceleromyograph designed to assess the degree of a neuromuscular block during anesthesia. The study compares the new three-dimensional technique with the established TOF Watch SX.

DETAILED DESCRIPTION:
The TOF 3D is a new acceleromyograph designed to assess the degree of a neuromuscular block during anesthesia. The study compares the new three-dimensional technique with the established TOF Watch SX. The time course of a neuromuscular block (onset, maximal block, time to recovery) is assessed simultaneously with both devices in 50 patients undergoing elective gynecologic surgery requiring neuromuscular block. The validity and reliability of the new technique is evaluated with a Bland-Altman- analysis.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing elective gynecologic surgery requiring general anesthesia and neuromuscular block

Exclusion Criteria:

* anticipated difficult airway
* Risk of pulmonary aspiration
* acute infection
* pregnancy
* renal or hepatic insufficiency
* neuromuscular disease
* chronic intake of drugs influencing neuromuscular block

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-08-31 (Actual); Primary Completion 2022-08-31 (Estimated); Study Completion 2022-08-31 (Estimated)

PRIMARY OUTCOMES:
TOF-R 90% | 12 months
  Difference of the 90% train-of-four (TOF) recovery time between both devices

SECONDARY OUTCOMES:
repeatability (precision) | 12 months
  Variance of 10 consecutive measurements around a linear regression line for each device
bias and limits of agreement (Bland-Altman analysis) | 12 months
  Difference between both devices against the average of both measurements (bias +- 2SD)

CONTACTS AND LOCATIONS:
Locations (1):
- KKH Dormagen, Dormagen, Germany

IPD SHARING:
Plan to Share IPD: No